CLINICAL TRIAL: NCT04253132
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Tolfenamic Acid for the Treatment of Progressive Supranuclear Palsy
Brief Title: Evaluation of Tolfenamic Acid in Individuals With PSP at 12-Weeks
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeuroTau, Inc. (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Zoltan Mari, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT 101-201
Record Dates: First submitted 2019-12-17; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — tolfenamic acid

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 50 mg daily oral dose (Active Comparator): 50 mg daily, oral dose of tolfenamic acid
  Interventions: Drug: Tolfenamic Acid
- 300 mg daily oral dose (Active Comparator): 300 mg daily, oral dose of tolfenamic acid
  Interventions: Drug: Tolfenamic Acid
- 600 mg daily oral dose (Active Comparator): 50 mg daily, oral dose of tolfenamic acid
  Interventions: Drug: Tolfenamic Acid
- Placebo control - 50 mg daily oral dose (Placebo Comparator): 50 mg daily oral placebo control
  Interventions: Drug: Placebos
- Placebo control - 300 mg daily oral dose (Placebo Comparator): 300 mg daily oral placebo control
  Interventions: Drug: Placebos
- Placebo control - 600 mg daily oral dose (Placebo Comparator): 600 mg daily oral placebo control
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tolfenamic Acid — Tolfenamic acid is an NSAID closely resembling mefenamic and flufenamic acid.
  Other Names: NT101
  Arms: 300 mg daily oral dose; 50 mg daily oral dose; 600 mg daily oral dose
Drug: Placebos — oral placebo
  Other Names: placebo
  Arms: Placebo control - 300 mg daily oral dose; Placebo control - 50 mg daily oral dose; Placebo control - 600 mg daily oral dose

SUMMARY:
This is a 12-week study of oral tolfenamic acid vs. placebo in Progressive Supranuclear Palsy (PSP)

DETAILED DESCRIPTION:
This is a 12-week, Phase 2a randomized, double-blind, placebo-controlled, parallel group study evaluating the safety and efficacy of tolfenamic acid (50 mg, 300 mg, and 600 mg daily) compared with placebo administered to subjects with PSP. The study will include 8 visits and a final telephone contact: screening (Week -6: Visit 1), randomization (7 to 10 days prior to Week 0: visit 2), treatment (Week 0 through Week 12: Visits 2 - 6), end of study Week 12: Visit 7), and telephone contact (Visit 8). Lumbar puncture will be obtained from consenting subjects at screening (Week -6: visit 10 and End of Study (Week 12: Visit 7) to primary exploratory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included in the study only if they meet all of the following criteria:

  * Probable or possible progressive supranuclear palsy defined as:
  * At least a 12-month history of postural instability or falls during the first 3 years that symptoms are present; and
  * At screening (Visit 1), a decreased downward saccade velocity defined as observable eye movement (deviation from the "main sequence" linear relationship between saccade amplitude and saccade velocity), or supranuclear ophthalmoplegia defined as 50% reduction in upward gaze or 30% reduction in downward gaze; and
  * Age at symptom onset of 40 to 85 years by history; and
  * An akinetic-rigid syndrome with prominent axial rigidity.
  * Aged 41 to 85 years at the time of screening (Visit 1).
  * Judged by investigator to be able to comply with neuropsychological evaluation at baseline and throughout the study.
  * Must have reliable caregiver accompany subject to all study visits. Caregiver must read, understand, and speak local language fluently to ensure comprehension of informed consent form and informant-based assessments of subject. Caregiver must also have frequent contact with subject (at least 3 hours per week at one time or at different times) and be willing to monitor study medication compliance and the subject's health and concomitant medications throughout the study.
  * Modified Hachinski score ≤ 3. This modified Hachinski will not include the focal neurological signs, symptoms or pseuodobulbar affect questions, given the prominence of all 3 in PSP.
  * Score ≥ 15 on the Mini-Mental State Examination (MMSE) at screening (Visit 1).
  * Written informed consent provided by subject (or legally-appointed representative, as appropriate) and caregiver (if not the legally-appointed representative) who are both fluent local language speakers.
  * Subject resides outside a skilled nursing facility or dementia care facility at the time of screening (Visit 1), and admission to such a facility is not planned. Residence in an assisted living facility is allowed.
  * If the subject is receiving levodopa/carbidopa, levodopa/benserazide, a dopamine agonist, catechol-o- methyltransferase (COMT) inhibitor, or other Parkinson's medication with the exception of Azilect (rasagiline), the dose must have been stable for at least 60 days prior to the screening visit (Visit 1) and must remain stable for the duration of the study. No such medication can be initiated during the study. Subjects receiving rasagiline or CoQ10 must be on a stable dose for at least 90 days prior to the screening visit (Visit 1).
  * Able to tolerate the MRI scan during screening with either no sedation or low dose lorazepam..
  * Able to ambulate independently or with assistance defined as the ability to take at least 5 steps with a walker (guarding is allowed provided there is no contact) or the ability to take at least 5 steps with the assistance of another person who can only have contact with one upper extremity.
  * Presence of symptoms for less than 5 years or the presence of symptoms for more than 5 years with a PSPRS baseline score ≥ 40.
  * Stable on other chronic medications for at least 30 days prior to screening.

Exclusion Criteria:

* Subjects will be excluded from the study for any of the following reasons:

  * Insufficient fluency in local language to complete neuropsychological and functional assessments.
  * A diagnosis of Amyotrophic Lateral Sclerosis (ALS) or other motor neuron disease.
  * Any of the following:
  * Abrupt onset of symptoms defined in inclusion criteria 1 associated with ictal events,
  * Head trauma related to onset of symptoms defined in inclusion criteria 1,
  * Severe amnesia within 6 months of the symptoms defined in inclusion criteria 1,
  * Cerebellar ataxia,
  * Choreoathetosis,
  * Early, symptomatic autonomic dysfunction, or
  * Tremor while at rest.
  * Presence of other significant neurological or psychiatric disorders including (but not limited to) Alzheimer's disease; dementia with Lewy bodies; prion disease; Parkinson's disease (which has not subsequently been revised to PSP), any psychotic disorder; severe bipolar or unipolar depression; seizure disorder; tumor or other space-occupying lesion; or history of stroke or head injury with loss of consciousness for at least 15 minutes within the past 20 years.
  * Within 4 weeks of screening (Visit 1) or during the course of the study, concurrent treatment with memantine; acetylcholinesterase inhibitors; antipsychotic agents (other than quetiapine) or mood stabilizers (e.g., valproate, lithium); or benzodiazepines (except as below).
  * Low dose lorazepam (not more than 2 mg) may be used for sedation prior to MRI scans for those subjects requiring sedation. Neuropsychological testing may not be performed after lorazepam administration.
  * Subjects who take short acting benzodiazepines (only temazepam or zolpidem are allowed) for sleep may continue to do so if they have been on a stable dose for 30 days prior to screening.
  * Clonazepam may be used for treatment of dystonia or painful rigidity associated with PSP if the dose has been stable for 90 days prior to screening and is not expected to change during the course of the study.
  * Treatment with lithium, methylene blue, tramiprosate, ketone bodies, latrepirdine, or any putative disease-modifying agent directed at tau within 90 days of screening (Visit 1).
  * A history of alcohol or substance abuse within 1 year prior to screening (Visit 1) and deemed to be clinically significant by the site investigator.
  * Any malignancy (other than non-metastatic dermatological conditions) within 5 years of the screening visit (Visit 1) or current clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease. For the non-cancer conditions, if the condition has been stable for at least the one year before the screening visit (Visit 1) and is judged by the site investigator not to interfere with the subject's participation in the study, the subject may be included.
  * Clinically significant laboratory abnormalities at screening(Visit 1), including creatinine ≥ 2.5 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of the normal reference range, vitamin B12 below the laboratory normal reference range, or thyroid stimulating hormone (TSH) above the laboratory normal reference range.
  * The systolic blood pressure measurement is > 190 or < 85 mm Hg. The diastolic blood pressure measurement is 105 or < 50 mm Hg at screening (Visit 1).
  * Abnormal ECG tracing at screening (Visit 1) and judged to be clinically significant by the site investigator.
  * Treatment with any investigational drugs or device within 90 days of screening (Visit 1).
  * Known history of serum or plasma progranulin level less than one standard deviation below the normal subject mean for the laboratory performing the assay.
  * Known presence of known disease-associated mutation in TDP-43, PGRN, CHMPB2 or VCP genes or any other frontotemporal lobar degeneration (FTLD) causative genes not associated with underlying tau pathology (e.g., Chromosome 9 associated FTD).
  * History of deep brain stimulator surgery other than sham surgery for deep brain stimulation (DBS) clinical trial.
  * History of early, prominent rapid eye movement (REM) sleep behavior disorder.
  * Women who are pregnant or lactating and women of childbearing potential who are not using at least two different forms of medically recognized and highly effective methods of birth control, resulting in a low failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
  * An employee or relative of an employee of the Sponsor, a clinical site, or contract research organization (CRO) participating in the study.
  * Significant anatomical nasal abnormality (e.g., septal deviation obstructing airflow to at least one nostril or septal perforation) or history of nasal turbinate surgery.
  * History of a clinically significant medical condition that would interfere with the subject's ability to comply with study instructions, would place the subject at increased risk, or might confound the interpretation of the study results.
  * Contraindication to the MRI examination for any reason (e.g., severe claustrophobia, ferromagnetic metal in body).
  * Structural abnormality on the MRI that precludes diagnosis of PSP, such as cortical infarct in brain region that might account for subject's symptoms.
  * In subjects receiving anti-Parkinson's Disease medication at the time of screening (Visit 1), in the opinion of the investigator substantial worsening of motor signs or symptoms compared with normal functioning following overnight withdrawal of the anti-Parkinson medication

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance of tolfenamic acid in individuals with PSP | 12-weeks
  Safety measures include: number of AEs, ECG changes, nasal examination and clinical laboratory tests

SECONDARY OUTCOMES:
CSF biomarker change from baseline | 12-weeks
  total tau, phosphporylated tau, amyloid beta peptide (1-42), NFL, ngrn, pNFH
Pharmacodynamic parameter of amyloid beta peptide | 12-weeks
  To measure treatment effect of tolfenamic acid in amyloid beta peptide concentrations in CSF
Pharmacodynamic parameter of total tau | 12-weeks
  To measure treatment effect of tolfenamic acid in total tau contcentrations in CSF
Pharmacodynamic parameter of phosphorylated tau | 12-weeks
  To measure treatment effect of tolfenamic acid in phosphorylated tau concentrations in CSF
Pharmacodynamic parameter of NFL | 12-weeks
  To measure treatment effect of tolfenamic acid in NFL concentrations in CSF
Pharmacodynamic parameter of ngrn | 12-weeks
  To measure treatment effect of tolfenamic acid in ngrn concentrations in CSF
Pharmacodynamic parameter of pNFH | 12-weeks
  To measure treatment effect of tolfenamic acid in pNFH concentrations in CSF concentrations

OTHER OUTCOMES:
Clinical global Impression of Change | 12-weeks
  Impression of change - CGI-C
Progressive Supranuclear Pallsy Rating Scale (PSPRS) | 12-weeks
  Change from baseline in disease severity. Higher values represent an increase in severity
Schwab and England Activities of Daily Living Scale (SEADL) | 12-weeks
  Change from baseline in ability to preform activities of daily living using a scale of 0 to 100 with 100 indicating total independance.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12-weeks
  Change from baseline measurement of cognitive function. Higher scores indicate better performance.
Phonemic Fluency | 12-weeks
  Change from baseline in Phonemic Fluency with higher score indicating a better health state
Color Trails Test | 12-weeks
  Change from baseline in Color Trails Test with lower score indicating a better. health state
Letter-number sequencing | 12-weeks
  Change from baseline in Letter-Number Sequencing with a higher score indicating a better health state
Clinical Global Impression of Disease Severity (CGI-ds) | 12-weeks
  Change from baseline in disease severity. Lower scores are associated with better health.
Geriatric Depression Scale (GDS) | 12-weeks
  Depression measurement of change from baseline with a higher score indicating depressive symptoms.
Plasma biomarkers | 12-weeks
  Tau, ngrn, NFL, pNFH, AB42

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Zawia, PhD, Study Director — NeuroTau, Inc.; Marwan Sabbagh, MD, Study Director — NeuroTau, Inc.
Locations (1):
- Lou Ruvo Center for Brain Health - Cleveland Clinic Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No